CLINICAL TRIAL: NCT02506270
Title: Effect of Airseal System Valve-less Trocar on the Ventilatory Parameters During Robotic-assisted Radical Cystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Ester Forastiere, Head of Department of Anaestesiology and Critical Care, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1/307.14
Record Dates: First submitted 2015-07-17; First posted 2015-07-23 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Mechanical Ventilation Pressure High

ARMS (2):
- AirSeal Trocar valveless (Active Comparator): patients are treated with the AirSeal-CO2-insufflator and trocar-system
  Interventions: Device: Airseal Trocar
- Conventional trocar (Sham Comparator): patients are treated with a conventional insufflation and trocar system
  Interventions: Device: conventional trocar

INTERVENTIONS:
Device: Airseal Trocar — 28 patients are treated with the AirSeal insufflation and trocar system
  Other Names: trocar valveless
  Arms: AirSeal Trocar valveless
Device: conventional trocar — 28 patients are treated with a conventional insufflation and trocar system
  Arms: Conventional trocar

SUMMARY:
The aim of the investigators' study is to investigate if the use of the AirSeal insufflation system impairs ventilatory parameters of patients less than a conventional system in patients undergoing robot-assisted laparoscopic cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for robotic-assisted Radical Cystectomy
* Written informed consent
* - ≥ 18 years of age

Exclusion Criteria:

* Patients who refuse participating in the study
* ejection fraction < 40%
* history of retinal vascular occlusion and ischaemic optic neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
change of dynamic compliance during surgery | 5min after induction,30min after trendelenburg position,1hours and 2hours after trendelenburg,30min and 1hour and 2hours after reduction Trendelenburg,5min after repositioning in supine position
  the variations of dynamic compliance during surgery are measured by mechanical ventilator and are expressed in ml/cmH2O

SECONDARY OUTCOMES:
change of peripheral oxygen saturation during surgery | 5min after induction,30min after trendelenburg position,1hours and 2hours after trendelenburg,30min and 1hour and 2hours after reduction Trendelenburg,5min after repositioning in supine position,1h after extubation
  the variations of peripheral oxygen saturation during surgery are measured by multiparameter patient monitor and are expressed in %
change of Peak Pressure during surgery | 5min after induction,30min after trendelenburg position,1hours and 2hours after trendelenburg,30min and 1hour and 2hours after reduction Trendelenburg,5min after repositioning in supine position
  the variations of peak pressure during surgery are measured by mechanical ventilator and are expressed in cmH2O

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena CI, Rome, Italy

REFERENCES:
- [Background] Herati AS, Andonian S, Rais-Bahrami S, Atalla MA, Srinivasan AK, Richstone L, Kavoussi LR. Use of the valveless trocar system reduces carbon dioxide absorption during laparoscopy when compared with standard trocars. Urology. 2011 May;77(5):1126-32. doi: 10.1016/j.urology.2010.06.052. Epub 2010 Oct 2. PMID 20888033